CLINICAL TRIAL: NCT02621255
Title: Effect of General and Regional Anesthesia on Fracture Healing
Brief Title: Effect of Anesthesia in Fracture Healing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Anesthesiologist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fracture Healing
Record Dates: First submitted 2015-11-26; First posted 2015-12-03 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Closed Fracture of Hip
MeSH Terms: interventions — Sevoflurane; Anesthesia, General; Bupivacaine; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia (Active Comparator): General Anesthesia: Effect of general anesthesia will compare with regional anesthesia without use of nonsteroid antiinflammatory drug usage. Propofol 2mg/kg and rocuronium will be administered to patients for anesthesia induction. Anesthesia maintenance will ensure with sevoflurane %2 and N2O/O2 %50/50 mixture.
  Interventions: Drug: Sevoflurane
- bupivacaine (Active Comparator): Regional Anesthesia: Effect of regional anesthesia will compare with general anesthesia without use of nonsteroid antiinflammatory drug usage. Combined epidural-spinal anesthesia will be performed to patients. %5 bupivacain and 20µg fentanyl will apply for spinal anesthesia. Anesthesia maintenance will ensure with bupivacain.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia type of performed for patient which has femur fracture.
  Other Names: general anesthesia
  Arms: General anesthesia
Drug: Bupivacaine — Anesthesia type of performed for patient which has femur fracture.
  Other Names: regional anesthesia
  Arms: bupivacaine

SUMMARY:
Investigator' s study designed to investigate effect of general and regional anesthesia on fracture healing.The 40 age and older ASAI-III patients who will operate due to femur fracture (except femur neck fracture) will be enrolled in this study after informed consent approval.

Subjects will be divided into two groups by a computerized randomization method. 40 patients will be enrolled in this study. General anesthesia will perform for 20 patients. Regional anesthesia will perform for 20 patients. Preoperative, 4. week and 12. weeks laboratory test which include blood and urine β-C terminal telopeptid (β-CTX), blood alkaline phosphatase and osteocalcin will test for all patients. All patients will not use nonsteroid anti-inflammatory drugs during study neither perioperative nor postoperative periods. fracture healing will be asses with clinical evaluation and laboratory tests.

DETAILED DESCRIPTION:
Investigator' s study designed to investigate effect of general and regional anesthesia on fracture healing.The 40 age and older ASAI-III patients who will operate due to femur fracture (except femur neck fracture) will be enrolled in this study after informed consent approval.

Subjects will be divided into two groups by a computerized randomization method. 40 patients will be enrolled in this study. Each group will have 20 patients. However a pilot study will perform for each groups with 10 patients. In Group G, all patients will be applied general anesthesia and 2 mg/kg propofol and 0,6 mg/kg rocuronium will administer to patients for induction of anesthesia. Maintenance of anesthesia will be made with %50-%50 O2/N2O and %2 sevoflurane. 0,1 mg/kg morphine will be held on last 10 minutes of operation for postoperative analgesia. Also, patient controlled analgesia with morphine(1 mg bolus and 20 min lockout time) will apply for postoperative analgesia. If it is necessary additional analgesic will provide with 100 mg peroral and intravenous tramadol. Regional anesthesia will perform for 20 patients which named Group R. In Group R combined epidural-spinal anesthesia will perform. Spinal %5 bupivacain 15 mg and 20µg fentanyl will apply and analgesia will provide with epidural bupivacain. Preoperative, 4. week and 12. weeks laboratory test which include blood and urine β-C terminal telopeptid (β-CTX), blood alkaline phosphatase and osteocalcin will all patients. All patients will not use nonsteroid antiinflammatory drugs during study neither perioperative nor postoperative periods. Fracture healing will be asses with clinical evaluation and laboratory tests. All measurements will be assessed with statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I-III
* Patients who will be operated for femur fracture
* 40 age and up patients

Exclusion Criteria:

* patients ASAIV and Up
* Haemodynamic unstable patients
* No patient's approval
* Femur neck fractures

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Bone turnover markers level-β-C terminal telopeptid (β-CTX) | up to 12 weeks
  Patients will follow until postoperative 12. weeks. β-C terminal telopeptid (β-CTX)(ng/mL or pg/mL) level will asses at preoperative, 4. week and 12. week

SECONDARY OUTCOMES:
Bone turnover markers level-osteocalcin | up to 12. weeks
  Patients will follow until postoperative 12. weeks.Osteocalcin (pg/mL) level will asses at preoperative, 4. week and 12. week
Bone turnover markers level-bone alkaline phosphatase | up to 12. weeks
  Patients will follow until postoperative 12. weeks.Bone alkaline phosphatase (U/L) level will asses at preoperative, 4. week and 12. week
Walking quality | up to 12. weeks
  Patients will follow until postoperative 12. weeks. Walking Quality will asses with clinical evaluation. With walker, with support( guided walk), full independent walk

CONTACTS AND LOCATIONS:
Overall Officials: Ersel Güleç, Principal Investigator — Cukurova University
Locations (1):
- Ebru Biricik, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obrant KJ, Ivaska KK, Gerdhem P, Alatalo SL, Pettersson K, Vaananen HK. Biochemical markers of bone turnover are influenced by recently sustained fracture. Bone. 2005 May;36(5):786-92. doi: 10.1016/j.bone.2005.02.009. Epub 2005 Mar 31. PMID 15804493
- [Background] Wolfl C, Schweppenhauser D, Guhring T, Takur C, Honer B, Kneser U, Grutzner PA, Kolios L. Characteristics of bone turnover in the long bone metaphysis fractured patients with normal or low Bone Mineral Density (BMD). PLoS One. 2014 May 1;9(5):e96058. doi: 10.1371/journal.pone.0096058. eCollection 2014. PMID 24788647
- [Background] Ikegami S, Kamimura M, Nakagawa H, Takahara K, Hashidate H, Uchiyama S, Kato H. Comparison in bone turnover markers during early healing of femoral neck fracture and trochanteric fracture in elderly patients. Orthop Rev (Pavia). 2009 Oct 10;1(2):e21. doi: 10.4081/or.2009.e21. PMID 21808683